CLINICAL TRIAL: NCT04134741
Title: Assessment of Effectiveness of Neuromuscular Training According to the Concept of Kinetic Control in Treatment of Lumbar Spine and Knee Pain and in Reduction of Risk of Injury in Female Football Players
Brief Title: Assessment of Effectiveness of Neuromuscular Training in Treatment of Lumbar Spine in Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: John Paul II University in Biała Podlaska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PopeJohnPaulIIStateSchHigherEd
Record Dates: First submitted 2019-09-25; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-09

CONDITIONS: Injury Leg; Back Pain; Sport Injury; Training Group, Sensitivity; Prevention
Keywords: prevention; back pain; soccer; football; female; sport injury; kinetic control
MeSH Terms: conditions — Leg Injuries; Back Pain; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: The players were placed at random in the studied groups, 9 participants in each group: A - group with additional Kinetic Control neuromuscular training; and B - group with standard training.
Who Masked: Investigator
Masking Description: None of the physiotherapists were personally involved in the preparation and the manner of performing the test.
  The random placement was performed with the use of computer software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinetic Control Group (Experimental): The players participated in the classic training and for 4 weeks (3 times a week) underwent the Kinetic Control neuromuscular training with assistance of a physical therapist.
  The duration of one training was 20-30 minutes.
  Interventions: Other: Kinetic Control
- Traditional Training Group (No Intervention): Players participated in the classic training.

INTERVENTIONS:
Other: Kinetic Control — The Kinetic Control training included a functional examination of motor disorders and individual training. The KC training included active exercises, active exercises with torso muscle resistance and exercises involving lower limbs.
  The duration of one training was 20-30 minutes.
  Other Names: Neuromuscular training
  Arms: Kinetic Control Group

SUMMARY:
The project aims to assess the effectiveness of neuromuscular training according to the concept of Kinetic Control (KC) in prevention and treatment of lumbar spine and knee pain and in reduction of risk of injury in female football players.

The study was designed as single-blind Randomized Controlled Trial (RCT) and conducted on a group of 18 female football players from University Club of the Academic Sports Association of Pope John Paul II State School of Higher Education in Biała Podlaska. Participants were randomly divided into two 9-person groups: A - used standard training and neuromuscular training (Kinetic Control) and B - used only standard training.

Main hypothesis:

The application of neuromuscular therapy (KC) reduces the risk of injuries and pain of the lumbar spine and the knee and improves the static and dynamic balance.

Research questions:

1. Will the application of the KC training reduce the risk and frequency of spine and knee injuries in females football players?
2. Will the KC training lead to reduction of the intensity of lumbar spine and knee pain?
3. Will the application of the KC training lead to increase in the torque strength of knee flexors and extensors and improved stability of the knee?
4. Will the application of the neuromuscular training (KC) lead to reduction of the disability level and improved functional level?

DETAILED DESCRIPTION:
The research was conducted upon acquiring an approval of the Bioethical Commission of Pope John Paul II State School of Higher Education in Biała Podlaska, no. 3/2018.

The study was designed as single-blind Randomized Controlled Trial (RCT) and conducted on a group of 18 female football players from University Club of the Academic Sports Association of Pope John Paul II State School of Higher Education in Biała Podlaska. Participants were randomly divided into two 9-person groups: A - used standard training and neuromuscular training (Kinetic Control) and B - used only standard training.

None of the physiotherapists were personally involved in the preparation and the manner of performing the test. Before commencing the tests, each participant was familiarised with their course, expressed their informed written consent for the participation and random assignment to the specified tested group.

The random placement was performed with the use of computer software.

The players participate in two training cycles over a year: from July to December and from January to June. Therefore, the above mentioned training regime will be performed twice.

A medical interview takes place before the training cycle. Physical examination, back pain functional scale (BPFS) and tests on the dynamographic platform will be performed two times - before and after each season.

ELIGIBILITY:
Inclusion Criteria:

* female players not taking nonsteroidal anti-inflammatory drugs (NSAIDs) for at least a week before the start of the study,
* written consent for the participation in the study.

Exclusion criteria:

* female players with acute inflammation (neuralgia) and massive intervertebral disk herniation requiring a surgery,
* female players who suffered from a lumbar spine and/or knee injury up to 6 months before the start of the study,
* female players with acute knee inflammation and after knee surgeries.

Ages: 19 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2019-06-16 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale of pain (VAS) | Visual analogue scale of pain (VAS) was carried out at the beginning of each season and after 6 months
  Visual analogue scale of pain (VAS) evaluates intensity of pain in the scale from 0 to 10. Maximum score means the highest level of pain.
Modified Laitinen's pain questionnaire | Modified Laitinen's pain questionnaire was carried out at the beginning of each season and after 6 months
  Laitinen's pain questionnaire took into account four indicators evaluated in the scale from 0 to 4: the intensity of pain, the frequency of its occurrence, the use of analgesic medications and limitation of the participant's motor activity. A research participant could have been granted from 0 to 16 points, the maximum score means the highest level of pain.
Stratford's back pain functional scale (BPFS) | Stratford's back pain functional scale (BPFS) was carried out at the beginning of each season and after 6 months
  In Stratford's scale (BFPS), the research participants assessed twelve actions related to everyday life activity in the scale from 0 to 5. The result fell within a range from 0 to 60 points, where the higher final result, the lower level of pain.

SECONDARY OUTCOMES:
Single leg small knee bend test | Single leg small knee bend test was carried out at the beginning of each season and after 6 months
  The test is performed in the standing position with feet a hip distance apart and parallel inner sides. The participant is then asked to transfer their body weight on one leg and raise the other leg over the ground. The body weight should be placed over the metatarsus. The participant is then asked to slightly bend the knee whilst keeping the heel on the ground. A photo is taken with a camera. Subsequently, computer software is used to determine the axis of the bent limb. The participant undergoes the test twice. If the test is not performed properly the first time, the participant is instructed how to perform the movement and the test is repeated.
  Proper test performance for the first time scores 2 points. Proper test performance after the guidance of the physical therapist scores 1 point and improper test performance twice scores 0 points.
Tests on the GAMMA dynamometric platform | Tests on the GAMMA dynamometric platform were carried out at the beginning of each season and after 6 months
  * Assessment of the load of lower limbs in the standing position for 30 seconds with eyes open. 1-1.15 was assumed as the proper load distribution ratio.
  * Assessment of the load of lower limbs in the standing position for 30 seconds with eyes closed. 1-1.15 was assumed as the proper load distribution ratio.
  * Assessment of the load of lower limbs in the squat test. The platform marks the load of lower limbs in three phases - standing up, stabilisation and squatting. 1-1.15 was assumed as the proper load distribution ratio in each phase.
  * Assessment of the load of lower limbs in the jumping test. The platform marks the load of lower limbs in three phases - jumping up, landing and stabilisation. 1-1.15 was assumed as the proper load distribution ratio in each phase.
Measurement of muscle force torque on a UPR-02A chair | Measurement of muscle force torque on a UPR-02A chair were carried out at the beginning of each season and after 6 months
  The test was performed under isometric conditions and included two measurements of each muscle group, for both the left and the right lower limb. The tested limb was stabilised at the 30-degree bend at the knee in order to measure the flexors and at the 60-degree bend in order to measure the extensors, assuming the 0 degree angle as full extension at the knee. In addition, the torso and distal thighs were stabilised with a belt. During the test, upper limbs were crossed on the chest. The axis of the torque measuring device was placed at the level of the knee joint gap (joint rotation axis). The measurements were taken in the following sequence: extension of the right limb, flexion of the right limb, extension of the left limb and flexion of the left limb.

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Zaworski, PhD, Study Director — John Paul II University in Biała Podlaska; Anna Kręgiel, PhD, Principal Investigator — John Paul II University in Biała Podlaska; Krystyna Gawlik, PhD, Study Chair — John Paul II University in Biała Podlaska; Joanna Baj-Korpak, PhD, Principal Investigator — John Paul II University in Biała Podlaska
Locations (1):
- Pope John Paul II State School Of Higher Education in Biała Podlaska, Biała Podlaska, Poland

IPD SHARING:
Plan to Share IPD: No